CLINICAL TRIAL: NCT06093698
Title: An Exploratory Study of A-337 in the Management of Malignant Solid Dose
Brief Title: An Exploratory Study of A-337 in the Management of Malignant Solid Dose Escalation and Expansion Phases
Acronym: A-337
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ITabMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-2021A
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Recurrent or Metastatic Solid Tumors
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): A-337dosage: 0.05, 0.15, 0.3, 0.6, 0.9, 1.2, 1.5 μg/kg/d
  Interventions: Biological: Recombinant Anti-EpCAM-CD3 Antibody Injection

INTERVENTIONS:
Biological: Recombinant Anti-EpCAM-CD3 Antibody Injection — Intravenous Infusion

SUMMARY:
Title: An Exploratory Study of A-337 in the Management of Malignant Solid Dose Escalation and Expansion Phases

DETAILED DESCRIPTION:
Protocol Number: IM-2021A Study Stage: Phase I Study Number: 2-3 sites Subject Number: up to 94 patients with recurrent or metastatic solid tumors, for whom there are no available effective standard treatments or for whom standard treatments have proven ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, all genders
* Patients with histologically or cytologically confirmed advanced malignant solid tumors who have failed standard treatment, have no standard treatment options, or are not suitable for standard treatment at this stage.
* The interval between the first dose of investigational drug and previous major surgery, medical device treatment, or local radiotherapy was at least 28 days. At least 21 days between the first dose of investigational drug and previous cytotoxic chemotherapy, immunotherapy, or biological agents; At least 14 days between he first dose of investigational drug and previous tumor-related endocrinotherapy and minor surgery; The interval between he first dose of investigational drug and small molecule targeted drugs was at least 21 days or 5 half-lives, whichever is longer; At least 14 days interval between the first dose of investigational drug and antineoplastic chinese traditional medicines.
* Patients with at least one measurable lesion on the basis of RECIST v1.1.
* ECOG ≤ 1
* Patients are willing to provide archival tumor tissue or undergo fresh tissue biopsy.
* Life expectancy is at least 3 months.
* Having adequate organ and bone marrow functional reserve, defined as follows:

  1. Blood routine (corrected with no growth factor support, blood transfusion, or other medication within 2 weeks before screening) ANC ≥ 1.5 ×109 /L,PLT≥ 75×109/L,HGB≥ 90 g/L
  2. hepatic parameters :TBIL ≤ 1.5 × ULN For patients with liver metastases or a history of Gilbert's syndrome/suspected disease,TBIL ≤ 3 ×ULN For patients without liver metastases,ALT≤ 2.5 ×ULN,AST≤ 2.5 ×ULN For patients with liver metastases,ALT or AST ≤ 5 ×ULN
  3. renal function:Cr≤ 1.5×ULN or CrCl≥ 45 mL/min (using The Cockcroft-Gault formula )
  4. coagulation function:APTT≤ 1.5 × ULN,INR≤ 1.5 × ULN. Patients who were in the therapeutic window for long-term use of anticoagulants who did not meet these criteria could be enrolled at the investigator's discretion.
* Participants are capable of providing written informed consent and adhering to the protocol.

Exclusion Criteria:

* Past or present malignant tumor diagnosed in the past 3 years and/or required treatment.Except for the completely resected basal and squamous cell skin cancers and any type in situ.
* Patients with CNS metastases, unless the metastases were treated and stable for at least 4 weeks and without taking systemic steroids ≥ 10 mg prednisone/day or equivalent.
* Patients suspected or confirmed immunocompromised:

  1. Patients with HIV
  2. Patients requiring systemic or local treatment with systemic steroids or any immunomodulatory drug (at a level that results in a systemic dose effect).E.g. High-dose oral or intravenous steroids > 10 mg/ day prednisone or its equivalent, or methotrexate > 15 mg once weekly).Allow topical, inhaled or topical use of steroids (at levels not thought to cause systemic dose effects);
  3. Patients with active autoimmune disease or a history of autoimmune disease with potential recurrence(e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autohemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).Exceptions are patients with type I diabetes, hypothyroidism that is manageable with hormone-replacement therapy, skin conditions (e.g., vitiligo, psoriasis, or alopecia) that require no systemic treatment, or childhood asthma/allergies that have resolved without any intervention in adulthood.
  4. Patients with allogeneic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation)
  5. Any other condition that was considered by the investigator to place the patient at unacceptable risk as a result of receiving immunomodulatory therapy.
* Anticancer therapy, including hormonal therapy, biological therapy, cellular therapy, or radiation therapy, was administered within 4 weeks prior to the initiation of study treatment, except in the following cases:

  1. Hormonal therapy for prostate cancer using gonadotropin-releasing hormone (GnRH) agonists.
  2. Hormone replacement therapy or oral contraceptives
* Participants with any disease, medical condition, or social factor that was judged by the investigator to be likely to affect the study results or adherence were excluded from the study according to the protocol:

  1. Uncontrolled acute infection or confirmed bacteremia.
  2. Patients with HIV or HBV,and HBV copy number > 1000/mL or HBV DNA titer > 200 IU/mL.And patients with HCV.
  3. Severe dyspnea, pulmonary insufficiency, or continuous oxygen therapy.
  4. The patients were classified as New York Heart Association (NYHA) class 3 or 4 or left ventricular ejection fraction (LVEF) < 50%.
  5. Myocardial infarction, unstable angina, stroke, or transient ischemic attack, or other cardiovascular events of grade III or higher, occurred within 6 months before dose administration.
  6. Severe arrhythmia or uncontrolled hypertension (systolic blood pressure > 180 mmHg and diastolic blood pressure > 100 mmHg) or diabetes mellitus.
* Patients with uncontrolled systemic infection.
* Patients with positive treponema pallidum antibody.
* Patients who had undergone major surgical procedures (craniotomy, thoracotomy, or laparotomy) or who had nonhealed wounds, ulcers, or fractures within 4 weeks before the administration of the first dose of investigational drug, with the exception of needle biopsy procedures.
* Patients with alcohol or drug dependence.
* Patients with mental disorders, including epilepsy or dementia, or poor adherence.
* Patients with tumor types of nonepithelial origin.
* Patients with received an EpCAM antibody class, CD3 dual antibody class, or CAR-T therapy.
* Patients who did not recover to grade 1 or less toxicity (CTCAE 5.0) from previous antineoplastic therapy(except alopecia) .Patients who did not recover to grade 1 or below (CTCAE 5.0) after radiotherapy (except no effect).
* Pregnant (positive pregnancy test), lactating women.Women of childbearing age who did not agree to use contraception for at least 3 months after signing the informed consent form until the end of the study.Women of childbearing age had a positive HCG test within 7 days before the first day of treatment.
* Male subjects who did not agree to use contraception for at least 3 months after signing the informed consent form until the end of the study (except surgical sterilization)
* Patients with a allergy to the study drug or its excipients.
* Patients who were deemed by the investigator to be ineligible for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Incidence and Characteristics of Adverse Events of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 1 (each cycle is 28 days)
  Incidence and characteristics of adverse events
Evaluate the MTD and DLT of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 1 (each cycle is 28 days)
  dose limited toxicity(DLT), maximum tolerance dose(MTD)

SECONDARY OUTCOMES:
Evaluate the PK(Cmax) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  Cmax
Evaluate the PK(Tmax) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  Tmax
Evaluate the PK（T1/2) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  T1/2
Evaluate the PK(Vd) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  Vd
Evaluate the PK(CL/F) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  CL/F
Evaluate the PK(MRT) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  MRT
Evaluate the PK(AUC) of A-337 in the Treatment of malignant Solid Tumors | At the end of Cycle 3 (each cycle is 28 days)
  AUC
Evaluate the efficacy evaluation（ORR） of A-337 in the Treatment of malignant Solid Tumors | At the end of each Cycle (each cycle is 28 days)
  ORR
Evaluate the efficacy evaluation（DCR） of A-337 in the Treatment of malignant Solid Tumors | At the end of each Cycle (each cycle is 28 days)
  DCR
Evaluate the efficacy evaluation（DDC） of A-337 in the Treatment of malignant Solid Tumors | At the end of each Cycle (each cycle is 28 days)
  DDC
Evaluate the efficacy evaluation（PFS） of A-337 in the Treatment of malignant Solid Tumors | At the end of each Cycle (each cycle is 28 days)
  PFS
Evaluate the efficacy evaluation（OS） of A-337 in the Treatment of malignant Solid Tumors | At the end of each Cycle (each cycle is 28 days)
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Qinghua Zhou, Doctor, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No